CLINICAL TRIAL: NCT03470844
Title: Using Cognitive Tests and Functional MRI to Investigate Long Term Cognitive Dysfunction Following a Critical Illness Due to a Major Burn Injury
Brief Title: Perioperative Research Into Memory: Cognitive Outcome Following Major Burns
Acronym: PRiMe
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); University of Westminster (Other)
Responsible Party: Principal Investigator, Marcela P. Vizcaychipi, Planned Care Surgery & Clinical Support Divisional Research Lead, Chelsea and Westminster NHS Foundation Trust
Other Study IDs: C&W13/099
Record Dates: First submitted 2016-05-10; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Major Injury
Keywords: Major burns; Intensive Care Medicine; Neurocognitive dysfunction; Functional magnetic resonance imaging; Neuroinflammation; Long term quality of life
MeSH Terms: conditions — Cognition Disorders; Neuroinflammatory Diseases | interventions — Patient Health Questionnaire; Diffusion Tensor Imaging; Spectrum Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 5-10 years post severe burn injury: Interventions:
  * Face-to-face neurocognitive tests examining attention, processing speed, working memory and executive function.
  * Psychological screening for the symptoms of depression, anxiety and post-traumatic stress disorder using the patient health questionnaire (PHQ9), generalised anxiety (GAD7) scoring systems and the trauma screening questionnaire.
  * fMRI studies including resting state fMRI, T1w-mpr, T2w-FLAIR, Diffusion Tensor Imaging (DTI) with 30 directions, Spectroscopy CSI chemical shift imaging, Spectroscopy SVS single voxel, susceptibility weighted imaging (SWI), double inversion recovery (DIR) and Perfusion ASL.
  * Quality of Life Self-Assessment data.
  Interventions: Behavioral: Face-to-face neurocognitive tests; Behavioral: Psychological screening; Other: fMRI; Behavioral: Quality of Life Self-Assessment data
- 2-5 years post severe burn injury: Interventions:
  * Face-to-face neurocognitive tests examining attention, processing speed, working memory and executive function.
  * Psychological screening for the symptoms of depression, anxiety and post-traumatic stress disorder using the patient health questionnaire (PHQ9), generalised anxiety (GAD7) scoring systems and the trauma screening questionnaire.
  * fMRI studies including resting state fMRI, T1w-mpr, T2w-FLAIR, Diffusion Tensor Imaging (DTI) with 30 directions, Spectroscopy CSI chemical shift imaging, Spectroscopy SVS single voxel, susceptibility weighted imaging (SWI), double inversion recovery (DIR) and Perfusion ASL.
  * Quality of Life Self-Assessment data.
  Interventions: Behavioral: Face-to-face neurocognitive tests; Behavioral: Psychological screening; Other: fMRI; Behavioral: Quality of Life Self-Assessment data
- 1-2 years post severe burn injury: Interventions:
  * Face-to-face neurocognitive tests examining attention, processing speed, working memory and executive function.
  * Psychological screening for the symptoms of depression, anxiety and post-traumatic stress disorder using the patient health questionnaire (PHQ9), generalised anxiety (GAD7) scoring systems and the trauma screening questionnaire.
  * fMRI studies including resting state fMRI, T1w-mpr, T2w-FLAIR, Diffusion Tensor Imaging (DTI) with 30 directions, Spectroscopy CSI chemical shift imaging, Spectroscopy SVS single voxel, susceptibility weighted imaging (SWI), double inversion recovery (DIR) and Perfusion ASL.
  * Quality of Life Self-Assessment data.
  Interventions: Behavioral: Face-to-face neurocognitive tests; Behavioral: Psychological screening; Other: fMRI; Behavioral: Quality of Life Self-Assessment data
- Control: Healthy age, gender, socioeconomic and educational level matched control.
  Interventions:
  * Face-to-face neurocognitive tests examining attention, processing speed, working memory and executive function.
  * Psychological screening for the symptoms of depression, anxiety and post-traumatic stress disorder using the patient health questionnaire (PHQ9), generalised anxiety (GAD7) scoring systems and the trauma screening questionnaire.
  * fMRI studies including resting state fMRI, T1w-mpr, T2w-FLAIR, Diffusion Tensor Imaging (DTI) with 30 directions, Spectroscopy CSI chemical shift imaging, Spectroscopy SVS single voxel, susceptibility weighted imaging (SWI), double inversion recovery (DIR) and Perfusion ASL.
  * Quality of Life Self-Assessment data.
  Interventions: Behavioral: Face-to-face neurocognitive tests; Behavioral: Psychological screening; Other: fMRI; Behavioral: Quality of Life Self-Assessment data

INTERVENTIONS:
Behavioral: Face-to-face neurocognitive tests — Assessment of attention, processing speed, working memory and executive function
  Other Names: - Hopkins Verbal Learning and Verbal Fluency tests; - CogState computerised battery
Behavioral: Psychological screening — Screening for the symptoms of depression, anxiety and post-traumatic stress disorder
  Other Names: - Patient health questionnaire (PHQ9); - Generalised anxiety (GAD7) scoring systems; - Trauma screening questionnaire
Other: fMRI — Brain volume, chemical markers, functional outcome
  Other Names: The functional MRI (fMRI) protocol includes:; - Resting state fMRI; - T1w-mpr, T2w-FLAIR; - Diffusion Tensor Imaging (DTI); - Spectroscopy; - Double inversion recovery (DIR) and Perfusion ASL
Behavioral: Quality of Life Self-Assessment data — EQ-5D will be converted into a utility score using standard EQ-5D UK tariffs
  Other Names: - EQ-5D

SUMMARY:
The long term survival of patients who require admission to critical care (CC) following a major burn injury (MBI) continues to improve with advanced clinical management. There has been increasing interest into cognitive dysfunction (CD) due to neuroinflammation (NI) following CC, anaesthesia, surgery, and the association of NI with diseases characterised by CD such as Alzheimer's disease. Patients who suffer a MBI and who subsequently require admission to CC will be at uniquely high risk for CD. MBI produces an exaggerated and prolonged systemic inflammatory response, with NI demonstrated in animal models. Additionally NI can be exaggerated by insults such as sepsis, anaesthesia, and surgical trauma, common and often necessary following MBI. The aim of this study is to identify CD using cognitive tests to examine for deficits in working memory and executive function. Test proposed to use are the Hopkins Verbal Learning and Verbal Fluency tests, and a validated computerised battery (CogState). Neuroinflammation and underlying pathophysiology using fMRI and spectroscopy, known to demonstrate biomarkers for CD and NI. QoL will be assessed using the validated EQ-5D tool.

The Inclusion criteria; patients who survive their burns injury (greater than 15% total body surface area) and require mechanical ventilation. Primary exclusion criteria; admission with toxic epidermal necrolysis syndrome, and evidence of head trauma.

DETAILED DESCRIPTION:
This is a novel, proof of principle, prospective, cohort design, observational clinical study to assess for functional brain reorganisation, structural changes and long-term cognitive dysfunction following major burns injury and intensive care admission. The hypothesis is that following a major burns injury and intensive care admission patients will have neurocognitive dysfunction and demonstrable functional alterations seen on functional MRI due to neuroinflammation as a result of the primary injury and subsequent inflammatory insults.

ELIGIBILITY:
Inclusion Criteria:

* Survival following admission to Chelsea and Westminster Burns Intensive Care Unit between 2004-2013 with a burn injury > 15% total body surface area, requiring intubation and ventilation

Exclusion Criteria:

* Patients under 16.
* Patients with toxic epidermal necrolysis syndrome or evidence of head trauma.
* Patients with evidence of risk to psychological safety from inclusion in study: any patient currently held under section of the Mental Health Act, any patient receiving formal psychiatric treatment (including involvement in a Personality Disorder Unit, being under voluntary section, current re-occurrence of chronic self harm), any patient currently detained at her Majesty's pleasure, any current substance abuse, or at the discretion of professional opinion following historical assessment of notes. - Patients with contraindications to MRI (patients with non-compatible pacemakers, patients with metallic foreign bodies e.g. metal sliver in their eye, patients with non-compatible surgical metal work, patients with severe claustrophobia).
* Patient refusal or inability to give full informed consent.
* Patients unable to understand plain verbal or written English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe burn injury admitted to a Burn Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function | 5 years
  Specifically to investigate cognitive tasks using a battery of computerised tests.

SECONDARY OUTCOMES:
Neuroinflammatory changes analysis. | 5 years
  Functional MRI scan

OTHER OUTCOMES:
Long-term quality of Life | 5 years
  EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Vizcaychipi, MD PhD FRCA, Study Chair — Chelsea and Westminster Hospital
Locations (1):
- The Burn Intensive Care Unit (BICU), Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No